CLINICAL TRIAL: NCT01841814
Title: Evolution of Bone Mineral Density (BMD) in Patients With Lymphoma Undergoing Chemotherapy: Prospective Longitudinal Study Over 12 Months.
Brief Title: Evolution of Bone Mineral Density (BMD) in Patients With Lymphoma Undergoing Chemotherapy
Acronym: LYMPHOS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: physician departure
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI11-DR-DAMAJ
Record Dates: First submitted 2013-04-22; First posted 2013-04-29 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Lymphoma; Osteoporosis
Keywords: Lymphoma; Osteoporosis; Chemotherapy; Patient with
MeSH Terms: conditions — Lymphoma; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lymphoma (Experimental)
  Interventions: Radiation: Bone densitometry.

INTERVENTIONS:
Radiation: Bone densitometry.

SUMMARY:
The purpose of this study is to assess changes of bone mineral density (BMD) at 12 months during the therapeutic management of patients with lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 80 with lymphoma,
* Histological diagnosis of Hodgkin's lymphoma (HL) or non-Hodgkin lymphoma (NHL) of follicular or aggressive (large cell or other),
* Patients who have not yet started their chemotherapy or who have started for less than a month
* Patient has signed informed consent.

Exclusion Criteria:

* Pathological fractures at the time of initial diagnosis of lymphoma,
* Compression of neurological epidural,
* Patients receiving treatment for osteoporosis (including bisphosphonates, selective modulators of estrogen receptor, calcitonin and parathyroid hormone Teriparatide).
* Discovery of osteoporosis or osteopenia fracture during the initial evaluation requiring the establishment of an osteoporosis treatment,
* Radiotherapy to the lumbar spine or hip studied,
* Location of bone lymphoma in the lumbar spine or hip studied,
* History of disorders affecting bone metabolism (prostate cancer with androgen, stomach cancer, hyperparathyroidism, hyperthyroidism, uncontrolled ...)
* A person incapable of giving consent personally,
* Pregnant or breastfeeding women,
* Protected Person (under guardianship)
* Patient not affiliated with a social security system.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Measurement of bone mineral density (BMD). | Change from Baseline of bone mineral density at 12 months.
  Patients will have a review of bone densitometry.

CONTACTS AND LOCATIONS:
Overall Officials: Gandhi DAMAJ, Doctor, Principal Investigator — CHU d'Amiens France
Locations (1):
- Gandhi DAMAJ, Amiens, Picardie, France